CLINICAL TRIAL: NCT02802462
Title: High-intensity Interval Training Enhances Mobilization/Functionality of Endothelial Progenitor Cells and Depressed Shedding of Vascular Endothelial Cells Undergoing Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jong-Shyan Wang, PhD, Rehabilitation Science, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 101-0408A3
Record Dates: First submitted 2016-05-19; First posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Hypoxia
Keywords: endothelial progenitor cell; hemodynamic; Exercise; HIIT
MeSH Terms: conditions — Hypoxia; Motor Activity

ARMS (3):
- High intensity-interval (HIT) (Experimental)
  Interventions: Behavioral: HIT
- moderate intensity-continuous (MCT) (Experimental)
  Interventions: Behavioral: MCT
- control (CTL) (No Intervention)

INTERVENTIONS:
Behavioral: HIT — 3-minute intervals at 40% and 80%VO 2max
  Arms: High intensity-interval (HIT)
Behavioral: MCT — sustained 60%VO 2max
  Arms: moderate intensity-continuous (MCT)

SUMMARY:
Exercise training improves endothelium-dependent vasodilation, whereas hypoxic stress causes vascular endothelial dysfunction. Monocyte- derived endothelial progenitor cells (Mon-EPCs) contribute to vascular repair process by differentiating into endothelial cells. This study investigates how high-intensity interval (HIT) and moderate intensity-continuous (MCT) exercise training affect circulating Mon-EPC levels and EPC functionality under hypoxic condition. Sixty healthy sedentary males were randomized to engage either HIT (3-minute intervals at 40% and 80%VO2max , n=20) or MCT (sustained 60%VO2max , n=20) for 30 minutes/day, 5 days/week for 6 weeks, or to a control group that did not received exercise intervention (n=20). Mon-EPC characteristics and EPC functionality under hypoxic exercise (HE, 100W under 12%O 2 ) were determined before and after various interventions.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary life
* Age 20~28

Exclusion Criteria:

* Smokers
* Users of medication/vitamins
* Any cardiopulmonary/hematological risk
* Regular exercise habits at least 1 year
* Exposed to high altitudes (>3000 m) for at least 1 year

Ages: 20 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Circulating progenitor cells conten | 6 weeks
  by flow cytometry before and after rehabilitation circulating progenitor cells conten before and after hypoxic exercise test

SECONDARY OUTCOMES:
Cardiopulmonary fitness | 6 weeks

OTHER OUTCOMES:
Cardiac hemodynamic measurement | 6 weeks
  evaluate cardiac hemodynamic response to exercise by noninvasive continuous cardiac output monitoring system
Cerebral hemodynamic measurement | 6 weeks
  Two pairs of near infrared probes were attached to each subject to monitor the absorption of near infrared light across left frontal cortex during graded exercise test
Muscular hemodynamic measurement | 6 weeks
  Two pairs of near infrared probes were attached to each subject to monitor the absorption of near infrared light across left vastus lateralis muscle during graded exercise test

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Shyan Wang, PhD, Principal Investigator — Chang Gung Memorial Hospital